CLINICAL TRIAL: NCT03673345
Title: Effect of Influenza Vaccination or Infection on the Development of Protective Immunity in Children
Brief Title: Development of Childhood Anti-Influenza Immunity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-0009; HHSN272201400005C; NCT03778203 (obsolete NCT alias)
Record Dates: First submitted 2018-08-30; First posted 2018-09-17 (Actual); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2021-03-29

CONDITIONS: Influenza; Influenza Immunisation
Keywords: B Cell; CD4 T Cell; Children; Influenza Vaccination; Protective Immunity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1A (Experimental): 0.25 mL dose of IIV-4 administered intramuscularly on days 0 and 28 of study year 1 and on day 0 of study year 2 in children 6-12 months of age who have not previously had an influenza infection or vaccination, n=20
  Interventions: Biological: Influenza Virus Quadrivalent Inactivated Vaccine
- Cohort 1B (Experimental): 0.25 mL dose of IIV-4 administered intramuscularly on day 0 of study year 2 after primary influenza infection in study year 1 in children 3-12 months of age, who have not previously had an influenza vaccination, n=20
  Interventions: Biological: Influenza Virus Quadrivalent Inactivated Vaccine
- Cohort 2A (Experimental): 0.25 mL (less than 36 months of age) or 0.5 mL (36 months of age or older) dose of IIV-4 administered intramuscularly on day 0 of study year 1 and day 0 of study year 2 in children greater than 12 months of age and born after 2009, who have previously received 2 doses of influenza vaccine prior to the study, n=60
  Interventions: Biological: Influenza Virus Quadrivalent Inactivated Vaccine
- Cohort 2B (Experimental): 0.25 mL (less than 36 months of age) or 0.5 mL (36 months of age or older) dose of IIV-4 administered intramuscularly on day 0 of study year 2 in children greater than 12 months of age and born after 2009, who have previously had an influenza infection in study year 1 and have received 2 doses of influenza vaccine prior to the study, n=20
  Interventions: Biological: Influenza Virus Quadrivalent Inactivated Vaccine
- Cohort 3A (Experimental): 0.5 mL dose of IIV-4 administered intramuscularly on day 0 of study year 1 and day 0 of study year 2 in children born between 2006 and 2009, who have previously received 2 doses of influenza vaccine prior to the study, n=30
  Interventions: Biological: Influenza Virus Quadrivalent Inactivated Vaccine
- Cohort 3B (Experimental): 0.5 mL dose of IIV-4 administered intramuscularly on day 0 of study year 2 in children born between 2006 and 2009, who have previously had an influenza infection in study year 1 and have received 2 doses of influenza vaccine prior to the study, n=20
  Interventions: Biological: Influenza Virus Quadrivalent Inactivated Vaccine
- Cohort 4A (Experimental): 0.5 mL dose of IIV-4 administered intramuscularly on day 0 of study year 1 and day 0 of study year 2 in children born between 2003 and 2006, who have previously received 2 doses of influenza vaccine prior to the study, n=30
  Interventions: Biological: Influenza Virus Quadrivalent Inactivated Vaccine
- Cohort 4B (Experimental): 0.5 mL does of IIV-4 administered intramuscularly on day 0 of study year 2 in children born between 2003 and 2006, who have previously had an influenza infection in study year 1 and have received 2 doses of influenza vaccine prior to the study, n=20
  Interventions: Biological: Influenza Virus Quadrivalent Inactivated Vaccine

INTERVENTIONS:
Biological: Influenza Virus Quadrivalent Inactivated Vaccine — A seasonal quadrivalent inactivated influenza vaccine (IIV4), prepared from influenza viruses propagated in embryonated chicken eggs, protecting against 2 influenza A subtypes (H1N1 and H3N3) and 2 influenza B subtypes (B Yamata lineage B Victoria lineage).

SUMMARY:
This study is a prospective surveillance of the immune response to seasonal vaccination in healthy children. The study will enroll a total of approximately 220 subjects. 140 children will be vaccinated with inactivated influenza vaccine (IIV) and will be divided into 4 age cohorts: 20 children between 6-12 months of age, 60 children greater than 12 months of age and born after 2009, 30 children with a birth date between 2006 and 2009, and 30 children with a birth date between 2003 and 2006. 80 children presenting with natural influenza infection prior to receipt of influenza vaccination also will be divided into 4 age cohorts: 20 children between 3-12 months of age, 20 children greater than 12 months of age with a birth date after 2009, 20 children with a birth date between 2006 and 2009, and 20 children with a birth date between 2003 and 2006. Influenza vaccines will be administered using age-appropriate guidelines in all years of the study: Fluzone 0.25 mL administered intramuscularly to children between 6 and 35 months of age and 0.5 mL to children 36 months of age and older. Subjects will be seen at one domestic site and their participation duration is 2 influenza seasons plus 1 optional season. The primary hypothesis being tested in this study is that there will be differences in the specificity, magnitude and functionality of CD4 T cell and B cell reactivity in a cohort of children depending on early childhood exposures. The primary objective of this study is to evaluate the relationship between influenza virus exposure, infection and vaccine history, and CD4 T cell reactivity in a cohort of children with well documented influenza exposures.

DETAILED DESCRIPTION:
This study is a prospective surveillance of the immune response to seasonal vaccination in healthy children. The study will enroll a total of approximately 220 subjects. 140 children will be vaccinated with inactivated influenza vaccine (IIV) and will be divided into 4 age cohorts: 20 children between 6-12 months of age, 60 children greater than 12 months of age and born after 2009, 30 children with a birth date between 2006 and 2009, and 30 children with a birth date between 2003 and 2006. 80 children presenting with natural influenza infection prior to receipt of influenza vaccination also will be divided into 4 age cohorts: 20 children between 3-12 months of age, 20 children greater than 12 months of age with a birth date after 2009, 20 children with a birth date between 2006 and 2009, and 20 children with a birth date between 2003 and 2006. Influenza vaccines will be administered using age-appropriate guidelines in all years of the study: Fluzone 0.25 mL administered intramuscularly to children between 6 and 35 months of age and 0.5 mL to children 36 months of age and older. Subjects will be seen at one domestic site and their participation duration is 2 influenza seasons plus 1 optional season. The primary hypothesis being tested in this study is that there will be differences in the specificity, magnitude and functionality of CD4 T cell and B cell reactivity in a cohort of children depending on early childhood exposures. The primary objective of this study is to evaluate the relationship between influenza virus exposure, infection and vaccine history, and CD4 T cell reactivity in a cohort of children with well documented influenza exposures.

ELIGIBILITY:
Inclusion Criteria:

1. Age:

   * Between 6 and 12 months at the time of enrollment to participate in the vaccination arm of age cohort 1A
   * Between 3 and 12 months at the time of enrollment to participate in the natural infection arm of age cohort 1B
   * > 12 months, birth date after 2009 for either the vaccination (A) or natural infection (B) arm of age cohort 2
   * Birth date between 2006 and 2009 for either the vaccination (A) or natural infection (B) arm of age cohort 3
   * Birth date between 2003 and 2006 for the vaccination (A) or natural infection (B) arm of age cohort 4
2. Gestational age of = / > 37 weeks at birth
3. Parent/Legally Authorized Representative (LAR) can provide informed consent, with children = / > 8 years of age providing informed assent
4. Available for the duration of the study
5. History of previous primary inactivated influenza vaccine (IIV) vaccination (at least 2 previous doses for age < 9 yrs, at least 1 previous dose for age 9 and older) only for participation in the vaccination (A) arm of age cohorts 2, 3, or 4
6. Acute illness documented by rapid influenza test, polymerase chain reaction (PCR) testing, or testing done by either University of Rochester Medical Center (URMC) Labs or Rochester General Hospital (RGH) Clinical Microbiology Labs to be due to influenza virus only for participation in the natural infection arms (B) of age cohorts 1-4
7. Children enrolled in the cohort A (vaccination cohort) are required to have an appropriate weight and vital signs as determined by a licensed medical provider. Children enrolled in the cohort B (natural infection cohort) are required to have an appropriate weight and clinically stable vital signs as determined by a licensed medical provider* *Children will not qualify for study participation if their weight is more than 2.5 standard deviations below population norms. This will be determined through calculation of a Z score using the PediTools website (https://www.peditools.org/) utilizing the appropriate Centers for Disease Control and Prevention (CDC) growth calculators for age

Exclusion Criteria:

1. Immunosuppression as a result of an underlying illness or condition (including the human immunodeficiency virus (HIV) or a primary immunodeficiency syndrome)
2. Active neoplastic disease
3. Use of potentially immunosuppressive medications currently or within the past year (including chemotherapeutic agents) or chronic (> 2 weeks) use of oral corticosteroid therapy
4. A diagnosis of asthma requiring chronic inhaled corticosteriod use
5. Participation in any clinical research study evaluating an investigational drug or therapy that is inconsistent with current standard of care within two (2) months of enrollment in this study
6. Previous administration of influenza vaccine in the current influenza season only for subjects in the vaccination arm (A) of the study (subjects presenting with acute influenza infection with vaccine failure will be eligible to enroll in the B cohorts)
7. Receipt of immunoglobulin or another blood product within the year prior to study enrollment
8. An acute illness within the previous 3 days or temperature > 38 degrees Celsius on screening except for participation in the natural infection (B) cohorts.
9. A contraindication to influenza vaccination except infants between 3 and 5 months presenting with natural influenza infection whose only contraindication is their current age.
10. Anemia in the previous 6 months (children on iron supplementation with no documentation of abnormal hemoglobin and/or hematocrit for >6 months will be allowed to participate in the study)
11. Recent (within 120 days) hospitalization, excluding hospitalization for delivery or subjects enrolled in the acute cohort who have been hospitalized for influenza-related reasons
12. Any medical history or other condition that the study Principal Investigator (PI) feels may have a more than a minimal impact on the immune response or may impact safety of the subject

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center - Strong Memorial Hospital - Infectious Diseases, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 2B | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B
Started | 5 | 3 | 57 | 12 | 21 | 7 | 20 | 0
Completed | 3 | 3 | 48 | 7 | 19 | 6 | 20 | 0
Not Completed | 2 | 0 | 9 | 5 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 3 | 3 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 4 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Unable to enroll in participants in Cohort 4B
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 2B | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B | Total
Number analyzed (Participants) | 5 | 3 | 57 | 12 | 21 | 7 | 20 | 0 | 125
Age, Continuous [Mean (Standard Deviation); unit: months] | 9.7 (1.6) | 7.2 (3.9) | 45.7 (25.7) | 39.5 (25.2) | 131.5 (15.3) | 130.9 (20.0) | 167.3 (9.1) |  | 81.4 (57.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 33 | 6 | 11 | 2 | 11 |  | 68
  Male | 1 | 2 | 24 | 6 | 10 | 5 | 9 |  | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 7 | 2 | 2 | 1 | 0 |  | 14
  Not Hispanic or Latino | 4 | 2 | 49 | 10 | 19 | 6 | 20 |  | 110
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 2 |  | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Black or African American | 2 | 0 | 13 | 5 | 1 | 0 | 1 |  | 22
  White | 2 | 2 | 32 | 3 | 11 | 7 | 15 |  | 72
  More than one race | 1 | 0 | 11 | 3 | 8 | 0 | 2 |  | 25
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 0 | 0 | 0 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Frequency of CD4 T Cells With a Given Functional Potential
Description: Percent of ICOS/PD1+ expressing cells within CXCR5+ CD4 T cell population
Time Frame: Year 2 (Visit 5)
Population: Unable to enroll participants into Cohort 4B
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 2B | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B
Number analyzed (Participants) | 2 | 3 | 42 | 6 | 18 | 6 | 17 | 0
Percentage | 0.70 (0.24) | 0.55 (0.31) | 0.52 (0.32) | 0.38 (0.27) | 0.40 (0.37) | 0.34 (0.17) | 0.30 (0.13) |

ADVERSE EVENTS:
Time Frame: 2 years
Description: AEs and SAEs not collected
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2A | Cohort 2B | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3 | 0/57 | 0/12 | 0/21 | 0/7 | 0/20 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT03673345/Prot_SAP_000.pdf